CLINICAL TRIAL: NCT03068286
Title: Tailored Internet-delivered Cognitive Behavioural Therapy for Depression and Anxiety in Patients With a Long-term Condition (Chronic Pain, COPD and Diabetes).
Brief Title: iCBT for Long-term Conditions in IAPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues
Sponsor: Derek Richards (Other)
Responsible Party: Sponsor-Investigator, Derek Richards, Director of Clinical Research and Innovation, Silver Cloud Health
Organization: Silver Cloud Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAPTLTC
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Chronic Pain; COPD; CHD - Coronary Heart Disease; Depression; Anxiety
MeSH Terms: conditions — Diabetes Mellitus; Chronic Pain; Pulmonary Disease, Chronic Obstructive; Coronary Artery Disease; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Space in Diabetes (Experimental): The SilverCloud interventions comprise of 8 modules of evidence-based CBT which have been tailored. Psychoeducational content in the diabetes programme focusses on the impact that mood can have on self-management and self-care when living with diabetes.
  Interventions: Behavioral: Space in Diabetes
- Space in COPD (Experimental): The SilverCloud interventions comprise of 8 modules of evidence-based CBT which have been tailored. Additional content on panic has been included in the COPD programme. Symptoms of COPD and anxiety can be closely linked, and this content provides CBT-based strategies for dealing with symptoms of panic and anxiety.
  Interventions: Behavioral: Space in COPD
- Space in Chronic Pain (Experimental): The SilverCloud interventions comprise of 8 modules of evidence-based CBT which have been tailored. A module on health anxiety, titled "Anxiety and your Health", has been added to the chronic pain programme. This module provides psychoeducational content on health anxiety, the unhelpful behaviours that accompany it and how these can negatively impact on the experience of pain.
  Interventions: Behavioral: Space in Chronic Pain

INTERVENTIONS:
Behavioral: Space in Diabetes — The SilverCloud interventions comprise of 8 modules of evidence-based CBT which have been tailored. Psychoeducational content in the diabetes programme focusses on the impact that mood can have on self-management and self-care when living with diabetes.
  Arms: Space in Diabetes
Behavioral: Space in COPD — The SilverCloud interventions comprise of 8 modules of evidence-based CBT which have been tailored.Additional content on panic has been included in the COPD programme. Symptoms of COPD and anxiety can be closely linked, and this content provides CBT-based strategies for dealing with symptoms of panic and anxiety.
  Arms: Space in COPD
Behavioral: Space in Chronic Pain — The SilverCloud interventions comprise of 8 modules of evidence-based CBT which have been tailored. A module on health anxiety, titled "Anxiety and your Health", has been added to the chronic pain programme. This module provides psychoeducational content on health anxiety, the unhelpful behaviours that accompany it and how these can negatively impact on the experience of pain.
  Arms: Space in Chronic Pain

SUMMARY:
SilverCloud provides internet-delivered interventions for depression and anxiety in NHS Mental Health Services. The interventions have proved successful in the management of depression and anxiety for clients presenting to mental health services, with recovery rates exceeding the national standard. Recently SilverCloud has embarked on tailoring the interventions for patients with long-term conditions including COPD, pain and diabetes. The purpose of the customisation is to make the interventions more meaningful and relevant to patients with LTCs, but all the while having the same goal of addressing depression and anxiety disorders. In doing so it would be expected that individuals might be in a better position to effectively self-manage their LTC. The current study, therefore, seeks to assess the possible effectiveness of implementing customised internet-delivered interventions for depression and anxiety for people with long-term conditions presenting to NHS mental health services.

DETAILED DESCRIPTION:
iCBT is the delivery of a tailored structured cognitive and behaviour therapy based programme, with support, to individuals with mild to moderate symptoms of depression and anxiety. There is now a substantial body of research evidence that supports the efficacy and effectiveness of internet-delivered cognitive behaviour therapy for depression and anxiety (Richards & Richardson, 2012; Andersson and Cuijpers, 2009). Historically, a number of iCBT interventions have been used in clinical practice in IAPT services. However, they have often suffered from poor engagement and consequently poor clinical outcomes. More recent developments in the field have produced more robust technological platforms, where content is delivered through a variety of media that enhance productivity, increase engagement and produce better clinical outcomes. The SilverCloud intervention has been demonstrated to be a clinical effective evidence-based cognitive behavioural treatment option (Richards et al., 2015).

Chronic illnesses can have profound effects on well-being, functional capacity and quality of life. Psychological comorbidities with an LTC can further contribute to the distress that is caused by these symptoms. Patients with comorbid depression and anxiety disorders and a long-term condition are associated with significantly higher health care utilisation, poorer outcomes from treatment and increased costs of care (Moussavi et al., 2007; Naylor et al., 2012). The IAPT programme in the UK provides effective treatments for depression and anxiety but these have been underutilized by people with LTCs and partially this is due to an underrecognition; one reason for this has been the traditional precedence set on managing the physical aspects of any LTC and effectively paying little attention to psychological comorbidity (Coventry et al., 2011).

Several pathfinders sites are currently involved in providing psychological treatment for long-term conditions, but to date, results have been limited due to several factors, such as delays in commencing programmes and funding issues. To this extent, SilverCloud wishes to implement their tailored "Space from…" series of programmes for long-term conditions - chronic pain, COPD and Diabetes. The purpose of the tailoring is to make the interventions more meaningful and relevant to patients with LTCs, but all the while having the same goal of addressing depression and anxiety disorders. In doing so it would be expected that individuals might be in a better position to effectively self-manage their LTC. The current study, therefore, seeks to assess the clinical feasibility of implementing customised internet-delivered interventions for depression and anxiety for people with LTCS presenting to IAPT services.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* English language speakers
* Have capacity to consent
* Has a chronic condition (Diabetes, COPD, Chronic Pain) with comorbid depression and/or anxiety.
* Suitable for step 2 intervention in NHS IAPT Services.

Exclusion Criteria:

* Exceed cut-off score for risk in terms of self-harm on the screening questionnaires.
* Receiving an intervention (therapeutic or biological) that is not a part of treatment as usual, or another trial.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Depression (as measured by the Patient Health Questionnaire) | Weekly for up to 8 weeks
  The Patient Health Questionnaire-9 (PHQ-9;(Kroenke, Spitzer, & Williams, 2001; Spitzer, Kroenke, & Williams, 1999) is a self-report measure of depression that has been widely used in screening, primary care, and research. The PHQ-9 items reflect the diagnostic criteria for depression outlined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) (American Psychiatric Association [APA], 2000). Summary scores range from 0-27, where larger scores reflect a greater severity of depressive symptoms. The PHQ-9 has been found to discriminated well between depressed and non-depressed individuals using the clinical cut-off of total score ≥10, with good sensitivity (88.0%), specificity (88.0%) and reliability (.89) (Kroenke et al., 2001; Spitzer et al., 1999).
Anxiety (as measured by the 7 item Generalised Anxiety Disorder inventory) | Weekly for up to 8 weeks
  The Generalized Anxiety Disorder-7 (GAD-7; (Spitzer, Kroenke, Williams, & Löwe, 2006) GAD-7 comprises 7 items measuring symptoms and severity of GAD based on the DSM-IV diagnostic criteria for GAD. The GAD-7 has good internal consistency (α = .92) and good convergent validity with other anxiety scales (Spitzer et al., 2006). Higher scores indicate greater severity of symptoms. The GAD-7 has increasingly been used in large-scale studies as a generic measure of change in anxiety symptomatology, using a cut-off score of 8 (D. A. Richards & Suckling, 2009).

SECONDARY OUTCOMES:
Diabetes Distress (As measured by the Diabetes Distress Scale) | Baseline (week 0) and end of treatment (week 8)
  The Diabetes Distress Scale (DDS; Polonsky et al., 2005; Fisher et al., 2008) is a 17-item measure that focusses on 4 aspects of distress associated with diabetes: emotional burden, regimen distress, interpersonal distress and physician distress. The measure and its 4 subscales have demonstrated good internal consistency (α > .87) and convergent validity with the Center for Epidemiological Studies Depression Scale, meal planning, exerecise and total cholesterol (Polonsky et al., 2005).
Pain Acceptance (As measured by the Pain Acceptance Questionnaire - revised) | Baseline (week 0) and end of treatment (week 8)
  The Chronic Pain Acceptance Questionnaire (Revised) (CPAQ-R; McCracken, Vowles & Eccleston, 2004) is a 20 item measure used to assess acceptance of pain in chronic pain patients and contains two subscales - activity engagement and pain willingness. The measure has demonstrated good levels of internal consistency (α = .80)
Clinical COPD Symptoms (As measured by the Clinical COPD Questionnaire) | Baseline (week 0) and end of treatment (week 8)
  The Clinical COPD Questionnaire (CCQ; Reda et al., 2010; Molen et al., 2003) is a 10 item measure that incorporates three subscales - symptoms, functional state and mental state. Each item is graded on a 7-point likert scale, where lower scores are indicative of a better COPD health status. Internal consistency of the measure has been found to be good (α = .91) (Molen et al., 2003)
Quality of Life (As measured by the EuroQOL 5D5L) | Baseline (week 0) and end of treatment (week 8)
  The EuroQol 5D5L (EQ5D5L) (Herdman et al., 2011) is a measure of health-related quality of life. The first part of the measure consists of 5 self-report items measuring the domains of mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each item has a possible five responses, which rank in severity (no problems - extreme problems). From these results, a societal index can be obtained, allowing for further analysis. The second part of the measure records self-reported health state on a visual analogue scale (VAS), a vertical line where the best and worst imaginable health states score 100 and 0, respectively.
Work and Social Adjustment (as measured by the Work and Social Adjustment Scale) | Baseline (week 0) and end of treatment (week 8)
  Work and Social Adjustment (WASA; Mundt, Marks, Shear & Greist, 2002) is a simple, reliable and valid measure of impaired functioning. It is a simple and reliable (α >.75) 5-item self-report measure which provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships.
Patient Experience (As measured by the Patient Experience Questionnaire) | End of treatment (week 8)
  The Patient Experience Questionnaire will be used to assess patient experience and satisfaction. This questionnaire forms a part of the IAPT minimum data set and is a national requirement in the UK. The PEQ contains several quantitative questions and open ended questions that are used to assess participant's views and satisfaction with service provision.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PD, Study Director — SilverCloud Health
Locations (1):
- Barnet, Enfield, and harringey Mental Health Trust, Enfield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richards D, Timulak L, O'Brien E, Hayes C, Vigano N, Sharry J, Doherty G. A randomized controlled trial of an internet-delivered treatment: Its potential as a low-intensity community intervention for adults with symptoms of depression. Behav Res Ther. 2015 Dec;75:20-31. doi: 10.1016/j.brat.2015.10.005. Epub 2015 Oct 21. PMID 26523885
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Moussavi S, Chatterji S, Verdes E, Tandon A, Patel V, Ustun B. Depression, chronic diseases, and decrements in health: results from the World Health Surveys. Lancet. 2007 Sep 8;370(9590):851-8. doi: 10.1016/S0140-6736(07)61415-9. PMID 17826170
- [Background] Naylor, C., Parsonage, M., McDaid, D., Knapp, M., Fossey, M., & Galea, A. (2012). Long-term conditions and mental health: the cost of co-morbidities. London, UK: The King's Fund.
- [Background] Coventry PA, Hays R, Dickens C, Bundy C, Garrett C, Cherrington A, Chew-Graham C. Talking about depression: a qualitative study of barriers to managing depression in people with long term conditions in primary care. BMC Fam Pract. 2011 Mar 22;12:10. doi: 10.1186/1471-2296-12-10. PMID 21426542
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Richards DA, Suckling R. Improving access to psychological therapies: phase IV prospective cohort study. Br J Clin Psychol. 2009 Nov;48(Pt 4):377-96. doi: 10.1348/014466509X405178. Epub 2009 Feb 9. PMID 19208291
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med. 2008 May-Jun;6(3):246-52. doi: 10.1370/afm.842. PMID 18474888
- [Background] McCracken, L. M., Vowels, K. E., & Eccleston, C. (2004). The chronic pain acceptance questionnaire. Pain, 107(1), 271-277.
- [Background] Reda AA, Kotz D, Kocks JW, Wesseling G, van Schayck CP. Reliability and validity of the clinical COPD questionniare and chronic respiratory questionnaire. Respir Med. 2010 Nov;104(11):1675-82. doi: 10.1016/j.rmed.2010.04.023. Epub 2010 Jun 11. PMID 20538445
- [Background] van der Molen T, Willemse BW, Schokker S, ten Hacken NH, Postma DS, Juniper EF. Development, validity and responsiveness of the Clinical COPD Questionnaire. Health Qual Life Outcomes. 2003 Apr 28;1:13. doi: 10.1186/1477-7525-1-13. PMID 12773199
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645